CLINICAL TRIAL: NCT05210959
Title: Reliability and Validity of the Turkish Version of the Affordances in the Home Environment for Motor Development-Infant Scale and Its Cultural Adaptation in Turkish Population
Brief Title: The Turkish Version of the Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS)
Acronym: AHEMD-IS
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Umut Apaydin, PhD, PT, Principal Investigator, Gazi University
Other Study IDs: 91610558-604.01.02.
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Premature; Infant Development; Environmental Exposure
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm or term born infants: Premature or term born infants between the aged 3-18 months were recruited in this study.
  Interventions: Other: The Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS)

INTERVENTIONS:
Other: The Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS) — The Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS) is an instrument that assesses the quality and quantity of motor development opportunities available in the home for infants aged 3 to 18 months. In this study, the Turkish version of the AHEMD-IS were constructed. Also, the validity and reliability of this version were examined.

SUMMARY:
The Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS) is an instrument that assesses the quality and quantity of motor development opportunities available in the home for infants aged 3 to 18 months. Since its initial publication, the AHEMD-IS has grown in popularity as a clinical tool and research criterion. Furthermore, the AHEMD-IS supports the claim that environmental factors can have a positive impact on future motor skills and later cognitive behaviors of infants. Also it is stated that environmental factors are associated with infant motor development and motor abilities. As of writing, it has been translated into eight languages from the original English version and has been reported as valid and reliable in countries such as China, Spain, Lebanon, and Persia. The aim of this study was to produce the Turkish version of the AHEMD-IS and to reveal the validity and reliability of this version.

DETAILED DESCRIPTION:
The International Classification of Health, Function, and Disability (ICF), developed by the World Health Organization, provides a standard framework for identifying the body functions and structures, activity restrictions, and difficulties in children's participation. One of the major innovations in the ICF is that it introduces an environmental factor classification that enables the identification of environmental barriers and facilitators for both the capacity and performance of activities and tasks in daily life. The physical, social, and behavioral environments in which humans live are shaped by environmental factors. Environmental factors are external to the individual and can have a positive or negative impact on an individual's participation, performance, and body function/structure.

One of the tools that evaluate the environmental home environment is the Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS). The AHEMD-IS is a valuable tool for assessing the home environment, one of the environmental factors affecting infant motor development, and is of considerable research and clinical importance. The importance of this questionnaire is based on evidence not just for the impact of the home environment on motor development, but also on future cognitive and social behaviors. Consequently, this study aimed to translate the original English version into Turkish and to test its psychometric properties for use in children aged 3-18 months. It was aimed to determine whether the translated questionnaire meets the appropriate and necessary standards for measuring the quantity and quality of motor competencies in the home environment of children aged 3-18 month.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-18 months

Exclusion Criteria:

* Children younger than 3 months or older than 18 months
* Congenital or systemic disease

Ages: 3 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study comprised of term and preterm newborns.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Affordances in the Home Environment for Motor Development (AHEMD-IS) | 2 weeks
  The AHEMD-IS is a questionnaire for assessing the home environment of children aged 3 to 18 months. The AHEMD-IS evaluates physical space (inside and outside), variety of stimulation and play materials (gross motor toys and fine motor toys). The scale consists of 41 items in total. For infants aged 3-12 months, the first 32 items are answered. It is stated that the other items are not suitable for babies under 12 months. All substances are applied to infants aged 12-18 months. Questions answered as yes or no are scored as 0 and 1 (0: no, 1: yes). Other questions are scored as 0, 1, 2, 3. For infants up to 12 months, a total of 66 points is obtained. For infants older than 12 months, a total of 93 points is obtained. A higher score indicates better environmental enrichment

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development -III (Bayley-III): | 2 weeks
  The Bayley-III is a widely used test battery to evaluate the cognitive, receptive, and expressive language, and gross and fine motor development in children aged 1-42 months. The cognitive scale in the Bayley-III test battery consists of 91 items. The receptive language scale consists of 49 items and the expressive language scale consists of 48 items. In the motor development section, the gross motor development scale consists of 72 items, and the fine motor development scale consists of 66 items. Items in each section are scored as 1 (can perform the desired skill) and 0 (cannot perform the desired skill). The raw scores obtained from all items are converted into scaled scores ranging from 1 to 19 points. Then, a composite score is obtained according to this scaled score. It is the composite score commonly used in studies. Composite scores range from 40 to 160. A higher score indicates better improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Bulent Elbasan, Prof., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cacola P, Gabbard C, Santos DC, Batistela AC. Development of the Affordances in the Home Environment for Motor Development-Infant Scale. Pediatr Int. 2011 Dec;53(6):820-5. doi: 10.1111/j.1442-200X.2011.03386.x. PMID 21507146
- [Background] Cacola PM, Gabbard C, Montebelo MI, Santos DC. Further Development and Validation of the Affordances in the Home Environment for Motor Development-Infant Scale (AHEMD-IS). Phys Ther. 2015 Jun;95(6):901-23. doi: 10.2522/ptj.20140011. Epub 2014 Dec 18. PMID 25524875
- [Background] Dinkel D, Snyder K, Cacola P. Affordances in the Home Environment for Motor Development-Infant Scale, Spanish Translation. Early Child Dev Care. 2019;189(5):802-810. doi: 10.1080/03004430.2017.1344653. Epub 2017 Jun 28. PMID 31217656
- [Background] Kavousipor S, Rassafiani M, Ebadi A, Solimani F, Hosseini A, Gabbard C. Cultural Adaptation and Psychometric Properties of the Persian Version of the Affordance in the Home Environment for Motor Development. Iran J Child Neurol. 2019 Winter;13(1):25-35. PMID 30598671